CLINICAL TRIAL: NCT01721213
Title: European Survey of Patient and Prescriber Understanding of Risks Associated With Trobalt™
Brief Title: Trobalt™ Products Risk Survey
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116771; WEUKBRE5744 (Other: GSK)
Record Dates: First submitted 2012-10-25; First posted 2012-11-05 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Epilepsy
Keywords: Epilepsy; survey; retigabine; patient information leaflet; physician's guide; Trobalt™
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients using Trobalt™: Use of Trobalt™ current use or at least one prescription filled within the previous three months.
  Interventions: Drug: Trobalt™
- Physicians prescribing AEDs: Physicians (neurologists) who prescribed AEDs at least once in the three months prior to the survey.
  Interventions: Drug: Trobalt™
- Physicians Prescribing Trobalt™: Physicians (neurologists) who have had experience of prescribing Trobalt™ specifically, from among those who have prescribed AEDs at least once in the three months prior to the survey.
  Interventions: Drug: Trobalt™

INTERVENTIONS:
Drug: Trobalt™ — Trobalt™ is a potassium channel opener used as an adjunctive treatment for partial onset seizures (a form of epilepsy where a seizure begins in a specific area in one side of the brain), with or without secondary generalization in adults aged 18 years and above with epilepsy.

SUMMARY:
As part of a European post-marketing commitment, GSK will conduct a survey of physicians' and patients' understanding of the significant risks associated with Trobalt™ (retigabine), as described in the Patient Information Leaflet (PIL) and the Physician's Guide. The goal of the surveys is to evaluate the effectiveness of the educational plan as specified in the European Risk Management Plan (RMP).

The objectives of this study are to assess patients' and prescribers' understanding and knowledge of the significant risks associated with Trobalt™ use as evaluated by a survey instrument.

This is a cross sectional survey of:

1. 250 patients recruited from across the following countries (United Kingdom, Sweden, Denmark, Switzerland, Spain, Slovakia and Norway) and up to 100 patients from Germany who are currently using or have filled a prescription for Trobalt™ at least once in the last 3 months.
2. 200 neurologists who have prescribed an anti-epileptic drug (AED) at least once in the last 3 months, and who were on the list to which a letter containing the Physician's Guide for Trobalt™ was distributed from across the following countries (United Kingdom, Sweden, Denmark, Switzerland, Spain, Slovakia and Norway). At least 75 of the neurologists will have prescribed Trobalt™. The survey will also aim to include up to 100 neurologists from Germany of which approximately 50 will have prescribed Trobalt™.

Patients eligible for the survey will be asked to take the survey online or via a telephone interview if the latter is preferred. Neurologists will be invited to take the survey online.

The selected countries were the first five countries to launch Trobalt™ (Germany, Denmark, United Kingdom, Switzerland and Sweden) and an additional three countries with launch in 2011, but with relatively high rates of uptake of Trobalt™ (Spain, Slovakia and Norway). The selection of countries includes Switzerland, which is not part of the European Union. However, the key messages regarding the risks with Trobalt™ are in alignment. The rationale for surveying the first five countries to launch is so that any issues identified from these countries regarding the effectiveness of the Physician's Guide and PIL in communicating the risks of Trobalt™ can be addressed as soon as possible, and the key messages can be revised in a timely manner. In addition, these countries are likely to provide the greatest number of neurologists with experience of prescribing Trobalt™, and their patients.

The primary outcome of the survey is the proportion of patients/neurologists providing correct responses to a series of questions concerning the significant risks associated with Trobalt™. The risks evaluated will be those described in the Trobalt™ PIL and in the Physician's Guide.

ELIGIBILITY:
Inclusion Criteria:

Patients will be required to meet all the following inclusion criteria:

* Use of Trobalt™: current use or at least one prescription filled within the previous three months.
* 18 years of age or older.
* Willing to take the online survey or have the survey administered via a telephone interview.

Physicians will be required to meet all the following inclusion criteria:

* Must have prescribed an AED at least once in the last 3 months
* Must be on the list to which the Physician's Guide for Trobalt™ was distributed.

Exclusion Criteria:

Patients meeting any of the following criteria will not be eligible to take the survey:

* Unable to understand and complete the survey by internet or phone.
* Currently an employee of GSK or UBC.

Physicians meeting any of the following criteria will not be eligible to take the survey:

- Currently an employee of GSK or UBC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A random sample of 350 patients who are currently being treated with Trobalt™or who have received Trobalt™within the last 3 months. Patients will be recruited by prescribers, who will be asked to provide survey invitations to their patients being treated with Trobalt™.
  A random sample of 300 neurologists prescribing anti-epileptic drug (AEDs) and who have been sent the Trobalt™ Physician's Guide. A sample of 200 neurologists will be recruited from across the same eight countries, with up to 100 neurologists from Germany. The recruitment will be from among those who have prescribed an AED at least once in the last 3 months, and who were on the list to which a letter including the Physician's Guide Trobalt™ was distributed. The survey will aim to recruit at least 75 physicians (from the seven specified countries) and 50 physicians from Germany with experience of prescribing Trobalt™ for sub-analyses, as these individuals would be expected to be more aware of the risks of Trobalt™.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The proportion of patients/neurologists providing correct responses to a series of questions concerning the significant risks associated with Trobalt™ The risks evaluated will be those described in the Trobalt™ PIL and in the Physician's Guide. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Ishihara L, Lewis A, Kolli S, Brickel N. European Survey of Prescriber Understanding of Risks Associated with Retigabine. Drugs Real World Outcomes. 2015;2(4):345-353. doi: 10.1007/s40801-015-0044-3. Epub 2015 Nov 16. PMID 26688787